CLINICAL TRIAL: NCT05248256
Title: Vertebral Bone Marrow in Lung Cancer Attention Trial (VMAT)
Brief Title: Vertebral Marrow Attention Trial (VMAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 21-0168; HSC20210892H (Other: UT Health San Antonio)
Record Dates: First submitted 2022-01-13; First posted 2022-02-21 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Dose Limitations to VMAT (Experimental): Patients confirmed to have T1-T3 N1-N3 (Stage IIIA-IIIC) or select Stage IV primary adeno- or squamous cell-carcinoma of the lung will be treated per standard of care; concurrent chemoradiotherapy for 6 to 6.5 weeks, followed by consolidative immunotherapy. A CT simulation scan is obtained with the patient in the treatment position allowing the radiation oncologist to delineate intended tumor targets and organs at risk (OAR). Using specialized treatment planning software, a radiation plan is generated with the goal of maximizing tumor coverage with intended prescription dose and minimizing unintended radiation dose to OARs below established thresholds. The primary intervention of this trial will be sparing the thoracic bone marrow. This will be done by delineating the thoracic bone marrow on the CT simulation scan and applying vertebral marrow-specific OAR constraints during treatment planning to optimally spare radiation dose to this structure during treatment
  Interventions: Other: Evidence-based radiation dose limitation to the vertebral bone marrow

INTERVENTIONS:
Other: Evidence-based radiation dose limitation to the vertebral bone marrow — The only intervention that will occur during the radiation treatment planning process will be the application of evidence-based radiation dose limitations to the vertebral bone marrow during treatment plan optimization in order to attempt to limit Grade 3 Lymphopenia (G3L) toxicity.

SUMMARY:
The purpose of this study is to see whether designing radiation to spare the vertebral bone marrow can limit the rates of lymphopenia during standard of care chemoradiation therapy and in the time to count recovery in the ensuing weeks. Secondary endpoints will examine whether this leads to improved disease control whether this is predictive of improved clinical outcomes such as rates of local recurrence (LR), metastasis free survival (MFS), overall survival (OS), and progression free survival (PFS) which will be followed prospectively up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 years
* Patients with AJCC (American Joint Committee on Cancer) 8 T1-T4, N1-N3, M0 stage IIIA-IIIC NSCLC (non small cell lung cancer)
* Patients with oligometastatic disease stage IV, M1 disease, in which definitive concurrent chemoradiotherapy to the thorax is planned
* CBC/CMP within these limits
* Absolute lymphocyte count>500/ml
* Hemoglobin>8 g/dL
* AST (aspartate aminotransferase)/ALT (alanine transaminase) <2.5 times of ULN
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* History of thoracic irradiation
* History of palliative radiation for the current malignancy under consideration
* Patients not being treated with definitive standard of care to the chest
* History of bone marrow disease and or leukemia
* History of prior cytotoxic chemotherapy for a disease other than for the current malignancy
* Polymetastatic disease, defined here as ≥3 or more extrathoracic metastases
* Administration of concurrent immunotherapy during radiation therapy, either as part of another clinical trial or otherwise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Limited G3L Toxicity | 6 weeks
  The primary end point will be evaluating whether implementing dosimetric constraints to the bone marrow will decrease rates of G3L toxicity in the peripheral blood compared to expected rates of 40% in large series examining toxicities during chemoradiation. Values will be expressed as a percentage rates of G3L lymphopenia.

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline to study end (up to 5 years)
  Overall Survival (OS), as measured from time of enrollment in the study
Progression free Survival (PFS) | Baseline to study end (up to 5 years)
  Progression Free Survival (PFS), either distant or local measured on routine surveillance imaging
Local Recurrence (LR) | Baseline to study end (up to 5 years)
  Local Recurrence (LR), measured per Response Evaluation Criteria in Solid Tumors (RECIST) criteria on routine imaging,
Metastasis Free Survival (MFS) | Baseline to study end (up to 5 years)
  Metastasis Free Survival (MFS), as measured on surveillance imaging
Change in Neutrophil to Lymphocyte ratio (NLR) | Baseline to study end (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Newman, MD, Principal Investigator — The University of Texas Health Science Center - Mays Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Service for Timely Access, Nashville, Tennessee
  - Mays Cancer Center, UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided